CLINICAL TRIAL: NCT06517251
Title: Aha BOOST Arm-hand BOOST Therapy to Enhance Recovery After Stroke: Clinical, Health Economic and Process Evaluation
Acronym: AHA-BOOST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Vrije Universiteit Brussel (Other); Jessa Hospital (Other); Revalidatieziekenhuis RevArte (Unknown); University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Prof Geert Verheyden, Professor Geert Verheyden, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S68329; T002323N (Other: FWO-TBM project)
Record Dates: First submitted 2024-07-03; First posted 2024-07-24 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: Randomized controlled trial; Upper extremity; Subacute stroke; Inpatient rehabilitation; Additional therapy; Clinical evaluation; Health-economic evaluation; Process evaluation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Assessor-blinded phase III randomized controlled trial with a parallel design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm-hand BOOST (Aha BOOST) (Experimental): Aha BOOST consist of 20 one-hour group sessions (spread over 4 weeks, 5 days a week) and one hour of individual therapy per week (divided in two times 30 minutes). This group will receive therapy for the upper extremity.
  Interventions: Other: Arm-hand BOOST
- Lower limb BOOST (L-BOOST) (Active Comparator): L-BOOST consist of 20 one-hour group sessions (spread over 4 weeks, 5 days a week) and one hour of individual therapy per week (divided in two times 30 minutes). This group will receive therapy for strengthening exercises the lower limbs and general reconditioning.
  Interventions: Other: Lower limb BOOST

INTERVENTIONS:
Other: Arm-hand BOOST — Aha BOOST consists of 20 one-hour BOOST sessions (spread over 4 weeks, 5 days a week) and one hour of individual technology-supported therapy per week (divided in two times 30 minutes), with the aim to provide intensive, goal-oriented upper limb therapy. The sessions will be executed with a maximum of two participants, under supervision of a trained therapist.
  The group sessions are focused on four key aspects: neurophysiology, sequences of reaching and grasping, de-weighting of the arm, and orientation of the hand towards objects. The different exercises are tailored to the individual patient, based upon ongoing assessment, discussion within the group of therapists, and individual treatment goals of the patient. Additionally, patients exercise two times 30 minutes per week with the AMADEO® (Tyromotion, Austria), an upper limb robotic device, focusing on finger and hand rehabilitation.
  Other Names: Aha BOOST
  Arms: Arm-hand BOOST (Aha BOOST)
Other: Lower limb BOOST — L-BOOST consists of 20 one-hour sessions and a personalized two times 30 minutes self-exercise program per week and focused on strengthening exercises for the lower limbs and general reconditioning. During the group sessions, circuit-class training is performed according to a standardized written protocol: 20 minutes of cycling on a sitting bike, 20 minutes of strengthening exercises for muscles around hip and knee (e.g. sit-to-stand training), 10 minutes of knee exercises using quadriceps bench in free swing mode and 10 minutes of leg press exercises. Again, a gradual increase in levels of difficulty is provided. Additionally, each patient receives a self-exercise program (balance; strengthening of foot, knee, and hip muscles; walking exercises), which is executed two times 30 minutes per week under minimal supervision of a therapist. None of the exercises involve the use of the upper limb.
  Other Names: L-BOOST
  Arms: Lower limb BOOST (L-BOOST)

SUMMARY:
The overall aim of this study is to establish the clinical- and cost-effectiveness of the arm-hand BOOST therapy when delivered on top of the usual care program in the sub-acute phase post stroke and to perform a process evaluation.

In this phase III RCT, 80 patients with stroke will be recruited from two inpatient stroke rehabilitation wards in Belgium and randomized to the experimental group receiving arm-hand BOOST therapy or the control group receiving the L-BOOST intervention, on top of their usual inpatient care program. The arm-hand BOOST program (1 hour/day, 5x/week, 4 weeks) consists of group exercises based on four key aspects, namely neurophysiology, sequences of reaching and grasping, de-weighting of the arm, and orientation of the hand towards objects. Additionally, technology-supported upper limb therapy will be provided two times 30 minutes per week. The L-BOOST intervention comprises a dose-matched program of lower limb exercises and general reconditioning. At baseline, after 4 weeks of training, 3 months after the intervention and at 12 months post stroke, outcome assessment will be performed. The primary outcome measure is the action research arm test (ARAT). Secondary outcomes include measures in the domain of upper limb function and capacity, independence, participation and quality of life. Multivariate ANOVA and sensitivity analyses will be used to compare change from baseline between groups. Information on medical costs will be collected to allow a health economic evaluation. Finally, a process evaluation will be performed to assist in identifying why arm-hand BOOST succeeds or fails unexpectedly or has unanticipated consequences, and how this can be optimized.

At the start of this study the investigators hypothesize that: (I) Aha BOOST will result in a significant greater improvement in arm-hand activity post-intervention, at follow-up and 12 months post stroke compared to control therapy (L-BOOST); (II) Aha BOOST will result in a significant greater improvement in upper limb function, performance, independence and activity of daily living, and participation post-intervention, at follow up and 12 months post stroke. (III) Investing in 24 hours of extra arm-hand therapy to subacute stroke patient in the inpatient rehabilitation setting can reduce the health-economic and societal cost 12 months post stroke.

DETAILED DESCRIPTION:
Data collection and transfer:

* Data will be collected by the clinical sites and by the external researchers from the KU Leuven, VUB and Jessa Hospital. Source documents will be used to collect the data, these can be on paper or digital document.
* Different kinds of data will be collected on paper, for example results of the clinical tests, questionnaires and diaries. A standardized case report form (CRF) will be completed during data collection, containing researchers notes, remarks concerning data quality, contextual information, deviations from the protocol, etc. These CRFs will be kept on paper, in the same folder as the research data that are collected on paper and will become part of the participant's source documentation. These forms will be digitalized by the researchers in the e-CRFs via REDCap. After digitalizing the data, these paper forms will be stored in a locked cabinet in the Department of Rehabilitation Sciences, Building The Nayer, of the KU Leuven. During data collection temporary storage is possible at building K on the health campus in Jette, of the VUB. Only authorized personnel will have access to this locked storage rooms as they will need to be granted access by the PI.
* The data collected by the clinical sites will consists of a combination of paper forms and digital documents. A ManGO platform (hosted by KU Leuven IT department) will be used for collecting these different pseudonymized data forms. The different paper forms and data received via ManGO will be processed to REDCap by the external researchers. After digitalizing the data, the paper forms will be stored in a locked cabinet in the Department of Rehabilitation Sciences, Building The Nayer, of the KU Leuven. During data collection temporary storage is possible at building K on the health campus in Jette, of the VUB. Only authorized personnel will have access to this locked storage rooms as they will need to be granted access by the PI. The recorded video's will be transferred via ZIVVER, after which they will processed by the external researchers and deleted both on the computer of the external researcher and in the clinical sites.
* Any participant records or datasets that are transferred to the Sponsor or any partners of the Sponsor will contain the study-specific participant identifier only; participant names or any information which would make the participant identifiable will not be transferred. All pseudonymized data relating to the Investigation must be transmitted in a secure manner to the Sponsor or any partners of the Sponsor via the ManGO platform or Zivver. Interim reports and a final report at the group level (without individual patient data) will be provided to the funder (FWO).

Power calculation:

* A power calculation was done based on the primary research question (evaluating the short-term clinical effect of Aha BOOST intervention versus the control intervention on arm-hand capacity). This give the following results: In the proof of concept RCT, an average difference of 7.8 points in ARAT between both groups, in change from pre- to post intervention was found. Furthermore, the standard deviation of change from pre- to post intervention was estimated to be 11.7 points for the ARAT scale. With 74 patients, the comparison between experimental and control group for change from pre- to post intervention will have 80% power to detect an average difference of at least 7.8 points at the 5% two-sided level of significance, assuming a standard deviation of at most 11.7 points.
* To account for an expected dropout of at most 8%, 80 patients will be recruited.

Statistical analysis:

1. Clinical data: Changes in ARAT-scores from baseline between patients in the experimental and control group will be compared. Change from baseline will be estimated in both groups based on a multivariate ANOVA model for the original ARAT scores, with time and treatment as main effects and with time by treatment interaction. As a further sensitivity analysis, the analysis will be repeated correcting for patient characteristics such as age, time post stroke, and cognitive impairments.

   Secondary outcome measures: Multivariate ANOVA and sensitivity analyses, as described above.

   Subgroup analyses: pre-specified subgroup analyses will be undertaken to explore the effects of the interventions in different types of stroke survivors, such as experiencing cognitive impairments, using appropriate caution about multiplicity in the interpretation of these results. If there appear to be different effects in different subgroups, this will be investigated using interaction or trend tests rather than the statistical significance of the result for the individual subgroup.
2. Health economic data: The economic evaluation will incorporate costs and health gains during the trial and follow-up period, adopting healthcare and societal perspectives. On the cost side, the evaluation will focus on the direct medical and non-medical costs, and on indirect costs depending on the perspective. The direct medical costs encompass all costs for treatment and follow-up from the healthcare perspective and all out-of-pocket contributions by the participant. Direct non-medical costs include transport costs, and home care help, whereas indirect costs include productivity loss (e.g. the number of days away from work). Productivity losses due to informal care will be documented and valued using the human capital approach. The effects are expressed in utilities, derived from the national values of the EQ-5D-5L.

   The cost-effectiveness of the intervention will be expressed in incremental cost per QALY (quality-adjusted life years), using a decision-analytic model based on the trial data with a time horizon of one year and on a lifetime horizon. The incremental cost per QALY will be calculated as a ratio of (Cost Experimental-Cost Control) / (Outcome Experimental-Outcome Control). The robustness of the results will be analyzed by probabilistic sensitivity analyses on the cost as well as on the outcome.

   Tornadodiagrams will be used to measure impact of individual components in healthcare utilization. Probabilistic sensitivity analyses by bootstrapping with replacement will be employed to test the robustness of the results, utilizing MS Excel, using a minimum of 1000 iterations to obtain 2.5% and 97.5% percentiles of the incremental cost-effectiveness ratio (ICER) distribution. In a second phase, the health economic model will be further extended from a one-year time horizon to a life-time horizon based on literature. A Markov-model is developed defining the health states in chronic stroke. Estimations on resource use and utilities for each health state are derived from international peer-reviewed literature. Special attention is paid to the transferability of the data to the Flemish healthcare context. This will done by validation checks within the research consortium and advisory board. Similar to the one-year model, probabilistic sensitivity analyses will be used to account for uncertainty around the input parameters
3. Process evaluation data: Qualitative data will be analyzed using content analysis (a deductive analysis based on the defined indicators) and thematic analysis (an inductive analysis where themes will be generated from the data by the researcher(s) using a generic qualitative approach). The aim is to interview +/- 16 interviewees to achieve meaning saturation per respondent group (patients, expert therapists and treating physicians). Approximately 48 interviews will be conducted, although the final numbers will be determined by saturation. Interviews will be audio recorded, transcribed at verbatim and analyzed in NVIVO. Different types of data-triangulation, by using different methods or data-sources to gain a more in depth understanding, will be applied: (1) methodological triangulation e.g. using a combination of interviews and observations; (2) data triangulation e.g. patients, Aha BOOST therapists and treating physicians; (3) theoretical triangulation e.g. involving researchers of different disciplines to look to the data from different perspectives; (4) investigator triangulation e.g. involving different researchers in data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Maximally 5 months after a first-ever unilateral, supra-tentorial stroke
* Minimally 18 years old
* A residual inpatient stay of minimally 4 weeks
* The ability to sit independently
* Motor impairment in the upper limb, as defined, based on the JSU diagram, as a score of 8-17 on stage 2 (synergies) of the Fugl-Meyer assessment upper extremity (FMA-UE) or a score of <8 on stage 2 of the FMA-UE, combined with a score of >6 on stage 5 (hand) of the FMA-UE.

Exclusion Criteria:

* Severe communication deficits as defined as a score of <24 out of 32 on the 'visual sentence comprehension' subscale of the Comprehensive Aphasia Test.
* Severe cognitive deficits as defined as a score of <18 out of 30 on the Montreal Cognitive Assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | Pre-intervention, immediate post-intervention (after 4 weeks of additional therapy), 3 months post-intervention and 12 months post-stroke.
  The Action Research Arm Test (ARAT) is the recommended outcome in stroke trials, measuring arm-hand capacity at ICF activity level.
  The total score ranges from 0 to 57, with higher scores representing better performance.

SECONDARY OUTCOMES:
Fugl-Meyer assessment- upper extremity (FMA-UE) | Pre-intervention, immediate post-intervention (after 4 weeks of additional therapy), 3 months post-intervention and 12 months post-stroke.
  Assessing the domain of upper limb function. The total score ranges from 0-66, where 0 indicates no motor function and 66 indicates intact motor function.
Stroke Upper Limb Capacity Scale (SULCS) | Pre-intervention, immediate post-intervention (after 4 weeks of additional therapy), 3 months post-intervention and 12 months post-stroke.
  Assessing the domain of upper limb capacity. The total score ranges from 0-10 and reflects the number of items a person can execute.
Barthel Index (BI) | Pre-intervention, immediate post-intervention (after 4 weeks of additional therapy), 3 months post-intervention and 12 months post-stroke.
  Assessing the domain of independence. The total score ranges from 0 (indicating total dependence) to 100 (indicating complete independence).
modified Rankin Scale (mRS) | Pre-intervention, immediate post-intervention (after 4 weeks of additional therapy), 3 months post-intervention and 12 months post-stroke.
  Assessing the domain of independence. mRS is a 7-point ordinal scale ranging from 0(no symptoms) to 6 (death).
Stroke Impact Scale (SIS) | Pre-intervention, immediate post-intervention (after 4 weeks of additional therapy), 3 months post-intervention and 12 months post-stroke.
  Assessing the domain of participation. For each subcategory, a domain score is calculated, ranging from 0 to 100, with higher scores indicating less impact.
EuroQOL (EQ-5D-5L) | Pre-intervention, immediate post-intervention (after 4 weeks of additional therapy), 3 months post-intervention and 12 months post-stroke.
  Assessing the domain of quality of life. This test compromises five dimensions, each scored on a 5-level scale: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems.

OTHER OUTCOMES:
Total of healthcare services that patients used from inclusion until 12 months post stroke. | From inclusion until 12 months post stroke.
  Following types of health care resource use will be documented and collected by the use of a diary and questionnaire: primary care visits, emergency visits, inpatient stays, outpatient services
Number and type of medication used by patients from inclusion until 12 months post stroke. | From inclusion until 12 months post stroke.
  The total number and type of medication used by the patients will be documented (number of days taken, dose, and frequency of intake). This data will be collected by using a diary.
The total of transport costs that patient had from inclusion until 12 months post stroke. | From inclusion until 12 months post stroke.
  The total transportation costs a patients incurs for their rehabilitation (including hospital visits, rehabilitation sessions,...) will be documented in a diary.
Total absence at work that patients experienced due to their stroke. | From inclusion until 12 months post stroke.
  Days away from work due to the stroke will be documented by using a questionnaire.
Number of home modifications that patients had to perform due to their stroke. | From inclusion until 12 months post stroke.
  The total number of home modifications that patients had to perform due to their stroke will be documented using a questionnaire.
Number of equipment and aids that patients have to use due to their stroke. | From inclusion until 12 months post stroke.
  The total number of equipment and aids that patients have to use due to their stroke will be documented using a questionnaire.
Socio-economic status of the participant | From inclusion until 12 months post stroke.
  The socio-economic status of the participant will be documented using a questionnaire, based on answers about income, education level, employment, and home situation.
Social benefits that participants receive from the government due to their stroke | From inclusion until 12 months post stroke.
  The social benefits participants receive from the government will be documented (e.g. sickness leave payments) by using a questionnaire.
Barriers and facilitators for implementation Aha BOOST in a rehabilitation center | Between first inclusion and 2 years after first inclusion.
  This outcome measure will be measured by performing interview with patients, treating therapists and the management involved in the implementation process. And by assembling communities op practice in which the Aha BOOST therapists can give feedback on the ongoing implementation process. The interviews with the patient will be performed immediately after their 4 weeks of Aha BOOST therapy. The interviews with the treating therapists and management will be conducted one year after the first included patient. The community of practices will be held frequently (couple of times a year, depending on the need expressed by the Aha BOOST therapists) and will be held for two years.
Content of study therapy a patient received (experimental or control therapy) | Between first inclusion and 2 years after first inclusion.
  The content of the study therapy will be collected by using therapy diaries. Those diaries will be collected during each therapy session for two years.
Content of usual care therapy a patient received | Between first inclusion and 2 years after first inclusion.
  The content of the usual care therapy will be collected by using therapy diaries. Those diaries will be collected during each therapy session for two years.
Quality of the Aha BOOST therapy | Between first inclusion and 2 years after first inclusion.
  The quality of the Aha BOOST therapy will be assessed by filming 2 therapy session of the Aha BOOST therapy per Aha BOOST patient. Observation schemes will be used to assess these videos on quality. These videos will be made during Aha BOOST therapy sessions for two years.

CONTACTS AND LOCATIONS:
Overall Officials: Verheyden Geert, Professor, Principal Investigator — KU Leuven
Locations (2):
- Belgium (2):
  - Revalidatieziekenhuis RevArte, Edegem, Antwerpen
  - Revalidatiecentrum K7 UZ Gent, Ghent, Oost-Vlaanderen

IPD SHARING:
Plan to Share IPD: Yes
Data will be available in a restricted access repository. The full pseudonymized dataset will be made available as open as possible, as closed as necessary after publication of the data. This because of the type of data (sensitive and personal).
  All the data will be made available for other research purposes regarding the same pathology (stroke) of the consortium partners (KU Leuven, VUB and Jessa), this after approval of an ethical committee.
  Additionally, the dataset could be made available for other doctors and institutions collaborating with the consortium partners after submitted a written request to the PI, approval of an ethical committee and based on a Data Transfer Agreement (DTA).
Time Frame: Data will be available upon publication of the research results, or as soon as possible thereafter.
Access Criteria: The data will be available via KU Leuven RDR. After publication of the results, the respective data will be made available via a suitable scientific repository, providing the necessary guarantees regarding GDPR compliance (i.e., KU Leuven repository, RDR). The dataset will be under restricted access.

REFERENCES:
- [Derived] Cornelis L, Cruycke L, Meyer S, De Smedt A, Fobelets M, Michielsen M, Vander Plaetse M, Putman K, Verheyden G. Additional arm-hand boost therapy (AHA-BOOST) in an inpatient rehabilitation setting during the subacute phase after stroke: protocol for a randomised controlled trial including a clinical, process and health economic evaluation. BMJ Open. 2025 Oct 10;15(10):e093079. doi: 10.1136/bmjopen-2024-093079. PMID 41073121
- See also: Project website — https://gbiomed.kuleuven.be/english/research/50000743/50000744/ahaboost/aha-boost-therapy